CLINICAL TRIAL: NCT00548366
Title: Comparison of Efficacy of 2 Gram Versus 4 Gram Sodium Restriction in the Management of Cirrhotic Ascites
Brief Title: Sodium Restriction in the Management of Cirrhotic Ascites
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Jennifer Cuthbert, UT Southwestern Medical Center at Dallas
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UTSouthwestern 062007-066
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Ascites
Keywords: cirrhosis; portal hypertension; ascites; sodium restriction
MeSH Terms: conditions — Ascites; Fibrosis; Hypertension, Portal | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4 gram sodium diet
  Interventions: Other: Sodium restriction
- 2 (Active Comparator): 2 gram sodium diet
  Interventions: Other: Sodium restriction

INTERVENTIONS:
Other: Sodium restriction — 4 gram sodium diet
  Other Names: No added salt diet
  Arms: 1
Other: Sodium restriction — 2 gram sodium diet
  Other Names: Low sodium diet
  Arms: 2

SUMMARY:
To determine the relationship between degree of sodium restriction and dietary compliance with clinical outcome of diuresis of portal hypertensive ascites in cirrhotic patients from a county hospital population.

Primary objective: Demonstrate that, when accompanied by the appropriate diuretic regimen, a No Added Salt diet (4 grams sodium per day) is as effective as a Low Sodium diet (2 grams sodium per day) in the management of cirrhotic ascites.

DETAILED DESCRIPTION:
Secondary objectives:

1. Demonstrate that patient acceptance is greater and diuresis faster with a No Added Salt diet compared with a Low Sodium diet
2. Demonstrate that side-effects of diuretic therapy are the same or less when patients are on a No Added Salt diet
3. Determine if glomerular filtration rate estimated from the modified diet in renal disease equation differs from that obtained by a 24 hour urinary creatinine in patients with cirrhotic ascites

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients of any etiology with ascites from portal hypertension diagnosed by paracentesis,
* Age 18-75
* Clinical or radiographic (abdominal CT or ultrasound) estimate of moderate - severe ascites
* Spanish-speaking subjects will be eligible for participation

Exclusion Criteria:

* Active drug or alcohol abuse,
* Active complications of SBP, hepatic encephalopathy, or GI bleed within 2 weeks,
* Hemorrhagic ascites, malignant ascites,
* Creatinine >2 mg/dL or CCl < 30 mL/min,
* K > 5.5 mmol/L,
* Diuretic refractory ascites
* Allergy to or intolerance of either spironolactone or furosemide
* Homelessness, incarceration, inability to follow up in clinic, or comply with diet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Control of ascites | 3 months

SECONDARY OUTCOMES:
Patient acceptance and compliance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Cuthbert, M.D., Study Director — UT Southwestern Medical Center at Dallas
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States